CLINICAL TRIAL: NCT03598478
Title: Tai Chi-muscle Power Training for Primary School Children With Developmental Coordination Disorder: A Randomized Controlled Trial
Brief Title: Tai Chi-muscle Power Training for Primary School Children With Developmental Coordination Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TC-MPT group (Experimental): Tai Chi-muscle power training group
  Interventions: Behavioral: TC-MPT
- TC group (Active Comparator): Tai Chi group
  Interventions: Behavioral: TC
- MPT group (Active Comparator): Muscle power training group
  Interventions: Behavioral: MPT
- Control group (No Intervention): Usual medical care is allowed.

INTERVENTIONS:
Behavioral: TC-MPT — Participants will receive two levels of training within each 90-minute session over a 12-week period: (1) TC training and (2) MPT. The TC training protocol consists of five basic TC movements. After receiving TC training, the participants in this group will take a 5-minute break and then receive MPT. During MPT, the participants will contract their major postural muscles bilaterally as fast as possible against a resistance equivalent to 70% of one repetition maximum.
  Arms: TC-MPT group
Behavioral: TC — Children in the TC group will skip the MPT session and practice TC movements repeatedly for 90 minutes. The exercise progression pattern in the TC-alone group will be the same as that in the TC-MPT group.
  Arms: TC group
Behavioral: MPT — Those children in the MPT group will perform strengthening exercises repeatedly for 90 minutes, with a short 5-minute break between the three sets of exercises if necessary. The exercise progression pattern in the MPT-alone group will be the same as that in the TC-MPT group.
  Arms: MPT group

SUMMARY:
Objectives: To compare the effectiveness of Tai Chi-muscle power training (TC-MPT), Tai Chi (TC) alone, muscle power training (MPT) alone, and usual care (as a control) for improving the limits of stability (LOS) of balance control in children with developmental coordination disorder (DCD) and to explore the relationship among LOS, falls, and functional performance in this population.

Design: A randomized controlled trial. Sample: 156 children with DCD. Interventions: TC-MPT, TC alone, MPT alone, or usual care for 12 weeks. Major outcomes: Outcomes will be evaluated at baseline, post-intervention, and a 3-month follow-up. An LOS test will give a dynamic LOS score, an isokinetic test will quantify leg muscle force production speed, Movement Assessment Battery for Children-2 will be used to assess functional motor performance, and fall history will be obtained via interviews.

Anticipated results and significance: The TC-MPT group is predicted to display the best LOS balance performance, which is associated with reduced fall incidents and improved functional performance. This novel training regime could be readily adopted into school or clinical settings to improve physical well-being in children with DCD, an outcome with positive socioeconomic implications.

DETAILED DESCRIPTION:
Children with developmental coordination disorder (DCD), who comprise about 6% of the primary school population, display marked movement and balance difficulties. Reduced limits of stability (LOS), the maximum spatial area in which a standing person can lean, in these children is a major concern because it predisposes them to falls and affects their motor development.

The investigator's recent studies demonstrate the underlying causes of impaired LOS in children with DCD to include suboptimal volitional control of the center of gravity (COG) and reduced leg muscle force production speed. Tai chi (TC) is a particularly suitable exercise for improving COG control, yet the speed of movement is too slow to improve muscle power. Hence, muscle power training (MPT), which can hasten leg muscle force production, in conjunction with TC (TC-MPT) may be an ideal therapy for improving LOS, preventing falls, and improving functional performance in children with DCD.

In the proposed study, the investigators will pioneer the treatment of both COG control and leg muscular deficit in children with DCD by incorporating MPT into TC. It is hypothesized that the LOS of balance control in these children can best be improved by treating both their COG control and muscular deficits. This hypothesis is supported by the prediction that TC-MPT is superior to either TC or MPT alone in improving LOS balance performance. Furthermore, improved LOS is associated with fewer fall incidents and better functional performance in children with DCD.

Objectives: To compare the effectiveness of TC-MPT, TC alone, MPT alone, and usual care (as a control) for improving the LOS of balance control in children with DCD and to explore the relationship among LOS, falls, and functional performance in this population.

Design: A randomized controlled trial. Sample: 156 children with DCD. Interventions: TC-MPT, TC alone, MPT alone, or usual care for 12 weeks. Major outcomes: Outcomes will be evaluated at baseline, post-intervention, and a 3-month follow-up. An LOS test will give a dynamic LOS score, an isokinetic test will quantify leg muscle force production speed, Movement Assessment Battery for Children-2 will be used to assess functional motor performance, and fall history will be obtained via interviews.

Anticipated results and significance: The TC-MPT group is predicted to display the best LOS balance performance, which is associated with reduced fall incidents and improved functional performance. This novel training regime could be readily adopted into school or clinical settings to improve physical well-being in children with DCD, an outcome with positive socioeconomic implications.

ELIGIBILITY:
Inclusion Criteria:

9- to 12-years-old

Classified as DCD according to the Diagnostic and Statistical Manual of Mental Disorders V (DSM-5)

A percentile score of < 5th percentile on the MABC-2

A total score of < 55 (for children aged 8 to 9 years 11 months) or < 57 (for children aged 10 or above) on the DCD questionnaire 2007 (Chinese version)

Attending a mainstream primary school (i.e., intelligence level within the normal range)

Exclusion Criteria:

Any known significant congenital, cognitive, psychiatric (other than comorbid attention deficit hyperactivity disorder [ADHD] or autism spectrum disorder [ASD]), neurological, sensory, musculoskeletal, or cardiopulmonary disorder that may affect motor performance

Receiving active treatment such as physiotherapy

Demonstrating excessive disruptive behavior during the assessments

Those unable to follow instructions properly

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of limits of stability | 0, 3, 6 months
  Computerized dynamic posturography - A dynamic limits of stability score (%), from 0-100%. A higher score represents a greater limits of stability (better).
Change of center of gravity control | 0, 3, 6 months
  Computerized dynamic posturography - time to complete the DLOS test (sec)

SECONDARY OUTCOMES:
Change of functional motor performance (raw data) | 0, 3, 6 months
  Movement Assessment Battery for Children-2 total test score
Change of functional motor performance (compared to norm) | 0, 3, 6 months
  Movement Assessment Battery for Children-2 total percentile rank (from 0-100 percentile). A higher percentile represents better functional motor performance.
Change of leg muscle force production speed | 0, 3, 6 months
  Isokinetic/ hand-held dynamometry: time taken to reach peak torque of the knee flexor and extensor muscles
Change of leg muscle strength | 0, 3, 6 months
  Isokinetic/ hand-held dynamometry: peak torque of the knee flexor and extensor muscles
Change of fall history | 0, 3, 6 months
  Self-reported and parent-reported falls

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Fong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided